CLINICAL TRIAL: NCT07125352
Title: Neutrophil to Lymphocyte Ratio in Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Marker of Severity and Prognosis
Brief Title: Neutrophil to Lymphocyte Ratio in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hieba gamal ezz-elragal awad, Assistant professor, Ain Shams University
Other Study IDs: FMASU R123/2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neutrophil lymphocyte ratio in COPD patients — Neutrophil lymphocyte ratio in determining severity and prognosis in exacerbation of COPD patients

SUMMARY:
Chronic obstructive pulmonary disease (COPD) stands as one of the leading causes of mortality worldwide. Acute exacerbations of COPD (AECOPD) lead to rapid respiratory function decline and worsened disease status. Despite recent studies, the ability of the neutrophil-to-lymphocyte ratio (NLR) to predict outcomes in patients with COPD remains controversial. It remains controversial whether NLR can predict clinical outcomes in hospitalized patients with AECOPD. Therefore, this study was conducted to investigate the predictive value of NLR for severity, adverse outcomes in hospitalized patients with AECOPD, and predicting treatment response in patients with AECOPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) stands as one of the leading causes of mortality worldwide, posing an increasing economic burden. Acute exacerbations of COPD (AECOPD) are defined as acute deterioration of respiratory symptoms requiring additional treatment, leading to rapid respiratory function decline, diminished quality of life, and worsened disease status. Neutrophils are the most common type of white blood cells (WBC) and participate in multiple inflammatory and immune processes through phagocytosis and cytokine release. Lymphocytes play a crucial role as coordinators of the inflammatory and immune processes in various physiological mechanisms. The neutrophil-to-lymphocyte ratio (NLR) is calculated by dividing the number of neutrophils by the number of lymphocytes in the peripheral blood test, reflecting an increase in neutrophils and a secondary decrease in lymphocyte count during the inflammatory response. The NLR is considered a biological marker reflecting the inflammatory condition and is increasingly recognized in various disorders such as pneumonia, malignant, coronary artery disease, or hematological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above, Patients who will be admitted at the Chest department, Ain-Shams University Hospitals, diagnosed with AECOPD based on the Global Initiative for Chronic Obstructive Lung Disease 2024 criteria

Exclusion Criteria:

* Patients who refused treatment.
* COPD patients with Malignancy, hematological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and above Patients who will be admitted at Chest department, Ain-Shams University Hospitals diagnosed with AECOPD based on the global initiative for chronic obstructive lung disease 2024 criteria
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The ratio of neutrophils to lymphocytes in (%) in the CBC | baseline
  investigate the relation between this % ratio and severity of symptoms and adverse hospitalization outcomes in hospitalized patients with AECOPD

SECONDARY OUTCOMES:
The ratio of neutrophils to lymphocytes in (%) in the CBC | 3 months
  - investigate the relation between this % ratio and spirometric indices (FEV1, FVC) as percent predicted in hospitalized patients with AECOPD in their follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasyea, Egypt